CLINICAL TRIAL: NCT06542055
Title: Comparison of the Effects of Preoperative Pulmonary Rehabilitation Exercises on Postoperative Anxiety and Muscle Strength in Lung Neoplasm Resection Patients
Brief Title: Compare the Effects of Preoperative Pulmonary Rehabilitation Exercises on Postoperative Anxiety and Muscle Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202207101RINC
Record Dates: First submitted 2023-02-13; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Lung Neoplasm
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative & postoperative exercise (Experimental): Will receive preoperative thoracic surgery health education manuals. Tailored preoperative pulmonary rehabilitation exercises and postoperative regular pulmonary rehabilitation exercises.
  Interventions: Other: Preoperative and postoperative pulmonary rehabilitation exercise
- Postoperative exercise (Active Comparator): Preoperatively, an education manual was provided; postoperatively, routine rehabilitation exercises were given.
  Interventions: Other: Preoperative education and postoperative exercise

INTERVENTIONS:
Other: Preoperative and postoperative pulmonary rehabilitation exercise — Besides receiving preoperative thoracic surgery health education manuals and postoperative regular pulmonary rehabilitation exercises, they also receive exercises originally tailored for pulmonary rehabilitation, including upper-body resistance exercise, lower-body resistance exercise, aerobic exercise, and respiratory muscle training for 4-7 days before surgery. In addition, a communication app group will be set up and an exercise diary will be provided.
  Arms: Preoperative & postoperative exercise
Other: Preoperative education and postoperative exercise — Receiving preoperative thoracic surgery health education manual and postoperative regular pulmonary rehabilitation exercises
  Arms: Postoperative exercise

SUMMARY:
Lung cancer, tracheal and bronchial cancers have long been the leading cause of cancer mortality in Taiwan. According to statistics, about 40% of newly diagnosed lung cancers are treated with surgery as the primary treatment. Although early surgery improves survival rates, most patients experience significant decreases in lung function, and physical function after surgery, which affects their quality of life.

Recent studies have found that preoperative and postoperative lung rehabilitation exercises play an increasingly important role in lung cancer care. In Taiwan, postoperative interventions for lung cancer have shown significant benefits, but there is a lack of evidence on the effectiveness of preoperative rehabilitation programs. To understand the effectiveness of the preoperative pulmonary rehabilitation program, a preoperative home rehabilitation program was designed to compare the efficacy of preoperative pulmonary rehabilitation in the current lung cancer care of patients undergoing lung neoplasm surgery.

DETAILED DESCRIPTION:
After confirming that the patient is eligible to participate and the patient signs a consent, basic information and The Hospital Anxiety and Depression Scale (HADS) will be completed at the preoperative clinic, and lung function tests, 30-second 30 seconds sit-to-stand test, grip strength test, physical status assessment, and activity level assessment will be performed. A healthcare instruction manual will be given at the preoperative clinic.

The preoperative exercise group (experimental group) and the control group will be assigned randomly. The preoperative exercise experiment group must complete the related exercises and records. The exercises include upper extremity resistance exercise, lower extremity resistance exercise, aerobic exercise, and respiratory muscle training.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing thoracic surgery with pulmonary resection (including wedge resection, segmentectomy, and lobectomy).
2. FEV1≦80%.
3. over 20 years old.
4. Those who can cooperate with pulmonary rehabilitation and sign the consent form.

Exclusion Criteria:

* Suspected metastases to other organs.
* Unsteady gait, limited mobility, unable to cooperate with exercise training
* Those who cannot communicate in Mandarin or Taiwanese.
* Oxygen saturation ≦85% at rest and without oxygen.
* New York Heart Association (NYHA) defines heart failure as grade IV.
* FEV1<30% and ever diagnosed COPD patients.
* S/P pneumonectomy patient.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Anxiety and depression | at preoperative OPD(baseline), admission, and discharge (through study completion, an average of 3 weeks)
  The patient's anxiety was assessed by the Hospital Anxiety and Depression Scale (HADS).
  The scale consists of 14 items, with 7 items for anxiety and 7 items for depression. The anxiety items are the odd-numbered questions, and the depression items are the even-numbered questions. Each item is scored on a four-point scale (0-3 points). The scores for the two subscales are calculated separately, each with a total score ranging from 0 to 21. Higher scores indicate greater levels of anxiety or depression.

SECONDARY OUTCOMES:
Lung function | Through preoperative intervention, rehabilitation exercises for the lungs were performed for up to 6 weeks after surgery until discharge. The time frame includes at baseline (preoperative outpatient department)、at admission and before discharge
  Lung function will be assessed using MicroLab Spirometer.
  1. Forced Vital Capacity；FVC (L)、(% predicted)
  2. Forced Expiratory Volume in First Second；FEV1)(L) 、(% predicted)
  3. Peak Expiratory Flow Rate；PERF(L/S)、(% predicted)
  4. FEV1/FVC(%)
Early Activity Level | Through preoperative intervention, rehabilitation exercises for the lungs were performed until about a month after surgery before discharge.The initial activity level after surgery (through study completion, an average of 3 weeks)
  ICCA (IntelliSpace Critical Care and Anesthesia) Ranges from 0-10, the higher level indicates better functional activity.
Grip strength | at preoperative OPD(baseline), admission, and discharge (through study completion, an average of 3 weeks)
  measured with TTM-YD digital grip strength dynamometer
Lower limb muscle strength | Through preoperative intervention, rehabilitation exercises for the lungs were performed until about a month after surgery before discharge.Time Frame at baseline(preoperative OPD).
  30 seconds sit and stand test
Physical condition | Through preoperative intervention, rehabilitation exercises for the lungs were performed until about a month after surgery before discharge.Time Frame at baseline(preoperative OPD)、the next day after surgery
  ECOG Performance Status Scale 0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng District, Taiwan

IPD SHARING:
Plan to Share IPD: No